CLINICAL TRIAL: NCT05874531
Title: End-expiratory Occlusion Test and Prediction of Preload Dependence: Echocardiographic and Hemodynamic Study in the ICU.
Brief Title: End-expiratory Occlusion Test and Prediction of Preload Dependence
Status: Completed | Type: Observational
Sponsor: Mongi Slim Hospital (Other)
Responsible Party: Principal Investigator, Mhamed Sami Mebazaa, Professor, Mongi Slim Hospital
Other Study IDs: TOTE Rea
Record Dates: First submitted 2023-04-28; First posted 2023-05-25 (Actual); Last update posted 2023-09-25 (Actual); Status verified 2023-09

CONDITIONS: Intensive Care Units; Ultrasonography; Blood Volume

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Responders to fluid challenge: Responders to fluid loading after an increase in sub-aortic VTI of more than 10% following a volume expansion.
  Interventions: Diagnostic Test: End-expiratory occlusion test
- Non responders to fluid challenge: Non responders to fluid loading after an increase in sub-aortic VTI of more than 10% following a volume expansion.
  Interventions: Diagnostic Test: End-expiratory occlusion test

INTERVENTIONS:
Diagnostic Test: End-expiratory occlusion test — 15 seconds end-expiratory occlusion

SUMMARY:
Three sets of measurements of hemodynamic parameters and sub-aortic VTI were performed: before and at the end of 15 seconds end-expiratory occlusion and after 250 mL saline administration over 10 minutes. Patients were considered responders to fluid loading after an increase in sub-aortic VTI of more than 10% following a volume expansion. SPSS was used for statistic study. A p < 0.05 was considered significant. The investigators performed univariate and then multivariate analysis.

DETAILED DESCRIPTION:
The patients included were in the supine position in a prone position at 30°. They had continuous monitoring by: electrocardioscopy; pulse oximetry and invasive blood pressure. Diuresis was monitored hourly.

A venous access to the superior vena cava territory (central venous catheter) was set up.

The patients were sedated with a Ramsay score > 4 and ventilated in controlled assisted mode.

The sub-aortic TVI (in cm) was measured in an apical 5-chamber section by pulsed Doppler using a 1-5 MHz ultrasound probe (M-Turbo sonosite). Three sets of measurements of hemodynamic parameters and sub-aortic VTI were performed: before and at the end of 15 seconds end-expiratory occlusion and after 250 mL saline administration over 10 minutes. At each point, the investigators noted the hemodynamic, ultrasound and biological parameters.

ELIGIBILITY:
Inclusion Criteria:

* Patients under mechanical ventilation and sedation in the intensive care units
* patients for whom the decision of 250 mL saline administration was taken for : hypotension (systolic pression under 90 mmHg or diatolic pression under 40 mmHg or tachycardia more than 90 pulse per minute or oliguria or the increase in cathecholamin needs.

Exclusion Criteria:

* Pulmonary Edema
* arrythmia
* dialysis
* Prone position

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Sixty patients were included. The main causes of admission in intensive care were traumatic causes, post operative care or medical causes. 35 were responders avec 25 non responders to fluid load.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2023-05-15 (Actual); Primary Completion 2023-08-15 (Actual); Study Completion 2023-09-15 (Actual)

PRIMARY OUTCOMES:
an increase in sub-aortic VTI of more than 10% | before and 10 minutes after 250 mL saline administration
  the variation of sub aortic VTI by cardiac ultrasonography

CONTACTS AND LOCATIONS:
Overall Officials: Mhamed Sami MS Mebazaa, Pr, Principal Investigator — Mongi Slim Hospital
Locations (1):
- Mongi Slim hospital, Tunis, Tunisia

IPD SHARING:
Plan to Share IPD: No